CLINICAL TRIAL: NCT06052865
Title: Serial Neuroimaging of Brain Injury and Brain Growth in the NICU in the Very Preterm Infant
Brief Title: Serial Brain MRI in Hospitalized Preterm Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: POM Wonderful LLC (Industry)
Responsible Party: Principal Investigator, Carmina Erdei, MD, Neonatologist, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019P003819
Record Dates: First submitted 2023-08-30; First posted 2023-09-25 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Preterm Birth Complication
Keywords: preterm; brain injury; neonatal rehabilitation
MeSH Terms: conditions — Premature Birth; Brain Injuries | interventions — Standard of Care; Intensive Care Units, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exposed: High neurological risk (Experimental): 25 very preterm infants with advanced neurological injury
  Interventions: Behavioral: SENSE-plus: The Supporting and Enhancing NICU Sensory Experiences 2nd Edition (SENSE II) program
- Exposed: Low neurological risk (Experimental): 25 very preterm infants with low/no neurological injury
  Interventions: Behavioral: SENSE: The Supporting and Enhancing NICU Sensory Experiences 2nd Edition (SENSE II) program
- Reference/ Standard of care (Other): 25 very preterm infants with no study exposure/ standard of care
  Interventions: Other: Reference/ Standard of care

INTERVENTIONS:
Behavioral: SENSE-plus: The Supporting and Enhancing NICU Sensory Experiences 2nd Edition (SENSE II) program — The SENSE II program was developed to engage parents in consistently providing positive, developmentally appropriate sensory exposures to their high-risk infants in the NICU every day of hospitalization. The SENSE II program includes specific doses and targeted timing (based on postmenstrual age) of evidence-based interventions of auditory, tactile, vestibular, kinesthetic, olfactory, and visual exposures to be conducted daily through hospitalization for preterm infants. Additionally, for very preterm infants with advanced neurological injury, additional 1-2 sessions of weekly motor therapy are added to the SENSE-II program
  Other Names: SENSE-plus
  Arms: Exposed: High neurological risk
Behavioral: SENSE: The Supporting and Enhancing NICU Sensory Experiences 2nd Edition (SENSE II) program — The SENSE II program was developed to engage parents in consistently providing positive, developmentally appropriate sensory exposures to their high-risk infants in the NICU every day of hospitalization. The SENSE II program includes specific doses and targeted timing (based on postmenstrual age) of evidence-based interventions of auditory, tactile, vestibular, kinesthetic, olfactory, and visual exposures to be conducted daily through hospitalization for preterm infants.
  Other Names: SENSE
  Arms: Exposed: Low neurological risk
Other: Reference/ Standard of care — Infants in the Unexposed group receive the NICU standard of developmental care throughout hospitalization.
  Other Names: NICU care
  Arms: Reference/ Standard of care

SUMMARY:
The purpose of this research study is to use serial magnetic resonance imaging (MRI) to define the timing and factors associated with brain injury as well as the pattern of brain growth of very preterm infants during hospitalization in the neonatal intensive care unit (NICU). In addition, the goal is to utilize early MRI to risk-stratify preterm infants and tailor rehabilitative interventions according to risk in order to explore associations between NICU rehabilitative intervention and short- and long-term outcomes of preterm infants.

DETAILED DESCRIPTION:
Neurological adverse outcomes of very preterm birth can range from severe, including cerebral palsy, hearing and vision impairments, language disorders and learning disability, to less severe, such as developmental coordination disorders, fine motor control deficits, and mild cognitive impairments. While there are numerous factors, such as birth weight, gestational age, interventricular hemorrhage, and bronchopulmonary dysplasia, that have been shown to be associated with neurobehavioral impairments, the underlying neural mechanisms leading to these impairments are not yet understood. In the unit where this study is conducted, the standard of care is that babies born extremely preterm, or those born very preterm with additional clinical risk generally undergo a term equivalent age magnetic resonance imaging (MRI). However, given the limited understanding of the etiology of many neuronal disorders particularly in preterm born infants, findings on these term MRIs can be presented to families with many unanswered questions in terms of causation and implication for future development.

The few previous studies undertaken to better understand the etiology of brain injuries have used longitudinal serial imaging of preterm infants' brain during their NICU stays to look at trajectories of brain structural growth and the development of brain injury. One study found profuse increases in cortical grey matter growth rates that were accompanied by decreases in relative unmyelinated white matter growth rates. Another study found that the most common term equivalent finding associated with preterm birth was diffuse white matter abnormality, although causation and factors associated with these growth alterations and injuries are yet to be fully understood. The main limitation of both serial imaging studies is the limited number of scans per patient that were performed. The average number of scans per infant for both studies was around 2, which often corresponded to one at birth and one at term equivalent age (prior to NICU discharge), and did not provide sufficient information to comprehensively characterize the pattern of brain growth and development in this population.

One study investigated the structure-function relationship in preterm infants between MRI and clinical measures of motor, neurological and neurobehavioral capacity. Researchers found strong associations between the General Movements Assessment, Hammersmith Neonatal Neurological Examination, NICU Neonatal Neurobehavioral Scale, Premie-Neuro, and Test of Infant Motor Performance that correlated with the early and term-equivalent MRI. Based on a review of 88 articles that evaluated sensory-based interventions integrated in the care of very preterm infants in the NICU, nurturing interventions were noted to correlate with improved infant development and lower rates of maternal stress.

One such evidence-based multisensory program for hospitalized preterm infants is the SENSE II Program: The Supporting and Enhancing NICU Sensory Experiences 2nd Edition (SENSE II). The SENSE II program was developed to engage parents in consistently providing positive, developmentally appropriate sensory exposures to high-risk infants in the NICU every day of hospitalization. The SENSE II program includes specific doses and targeted timing (based on postmenstrual age) of evidence-based interventions of auditory, tactile, vestibular, kinesthetic, olfactory, and visual exposures to be conducted daily through hospitalization for preterm infants. The program also comprises a curated collection of parent educational materials aimed at guiding parents on infant sensory development, parenting in the NICU, and coaches families how to tailor nurturing interventions contingently upon infant responses and tolerance.

While these previous studies using serial imaging techniques provide a great foundation to understand individual brain development in the preterm infant, the lack of systematic regular serial MRI scans over the course of the entire NICU stay leaves room for future investigations to define the timing and factors associated with brain injury, as well as the pattern of brain growth in the preterm infant over the course of NICU the hospitalization. Newer imaging analysis methods are now available that allow regional brain volumes to be studied, which was not previously possible. Also, transporting small infants out of the NICU to the MRI scanner was a major barrier to carrying out serial studies without risk. This can now be overcome by new in-NICU MRI scanning technologies. As such, the Aspect Embrace Neonatal MRI System is an FDA-approved device which uses innovative technology to safely and effectively image infants within the NICU care environment. This type of in-NICU MRI scanner is available at this study site, specifically designed for infant neuroimaging and featuring a built-in incubator, self-contained magnet, and continuous video monitoring.

The present study plans to enroll very preterm infants who will receive brain MRI scans approximately every 2 weeks from enrollment until term-equivalent age, with an anticipated total of at least 3 brain scans, to monitor brain growth and evolution of injury throughout NICU hospitalization. Exposed infants will be categorized into two exposure groups (group 1: low-risk, and group 2: high-risk) based on the degree of neurological injury detected on early brain magnetic resonance imaging at study enrollment. Infants in the exposure groups will be compared with a reference group (group 3: unexposed). The primary outcome of this study consists of characterization of brain growth and development among preterm infants receiving NICU-based neuropromotive interventions compared to preterm infants receiving the standard of care at term-equivalent. Secondary outcomes include measures of infant neurodevelopment and parent-reported infant and family functioning at NICU discharge and at two years of age.

ELIGIBILITY:
Inclusion

* currently admitted to the BWH NICU
* born before 33 weeks completed gestational age
* birth weight 0.5-4.5 kg
* is stable condition per clinical care team

Exclusion

* confirmed or suspected congenital anomaly or genetic syndrome
* congenital TORCH infection

Ages: 22 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-14 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of brain injury on term equivalent brain MRI in very preterm infants | 3 months, average length of hospitalization for very preterm born infants
  Term equivalent brain MRIs will be assessed to characterize brain injury, including elements of: white matter abnormalities, cortical gray matter abnormalities, deep gray matter abnormalities, and cerebellar abnormalities. A total (global) brain injury score will be calculated as the sum of regional brain abnormalities total scores, with higher scores indicating more advanced level of injury as per the established scoring system for hospitalized preterm infants published by Kidokoro et al. The score will reveal the following categories for brain injury: no injury (total score 0-3), mild injury (score 4-7), or moderate-severe injury (total score 8 or above).
Incidence and severity of white matter injury on early brain MRI before term-equivalent age for very preterm infants | 3 months, average length of hospitalization for very preterm born infants
  Enrolled infants will undergo at least 2 early brain MRIs before term-equivalent age during the NICU hospitalization. Presence or absence of white matter injury on early brain MRIs will be categorized as follows: normal (no white matter lesions), minimal (3 or fewer areas of T1 signal abnormality), or moderate-severe (> 3 areas of T1 signal abnormality)

SECONDARY OUTCOMES:
Standardized assessment of developmental performance across multiple areas (cognitive, language, motor) at 2 years corrected age | Up to 2 years corrected age
  General developmental skills will be assessed using the Bayley Scales of Infant and Toddler Development 4th Edition, which will be administered by a licensed clinical psychologist at 2 years corrected age. This assessment will provide standard scores and percentiles for each patient's performance in each of these domains: cognitive, language, motor. Scores will then be analyzed and presented as Average/Means and Standard Deviations for each study group, and performance among groups will be compared. For each of the Bayley assessment categories, the Average or Mean is considered to be 100, with a 1SD interval of 90-110, where higher scores represent better performance.
Parent-reported child developmental performance (optional parent questionnaire) | Up to 2 years corrected age
  Child developmental performance measures will be collected with parent questionnaires given to parents at discharge and in follow-up up at 2 years corrected age. This will be assessed using The Ages and Stages Questionnaire, using the age-appropriate version. The ASQ scores will be compared with published referenced norms for age as per the Ages and Stages Questionnaire manual. Scores in each subdomain range on a scale from 0 (minimum) to 60 (maximum), with higher scores representing better performance.
Parent-reported child risk for autism (optional parent questionnaire) | 2 years corrected age
  The Modified Checklist for Autism-Revised (M-CHAT R) in Toddlers is a parent-report questionnaire that screens for behaviors commonly found in children with Autism Spectrum Disorders. Scoring will be performed as per published American Academy of Pediatrics guidelines, with higher scores representing a higher risk for autism. The risk categories will be classified as follows: score of 0-2 (non-critical items): "Low risk"; score of 3-6: "Medium risk" (or ≥2 critical items on M-CHAT), and score of 8-20: "High risk".
Incidence of parental stress (optional parent questionnaire) | Up to child's 2 years corrected age
  The Parental Stress Scale (PSS) or Parental Stress Scale (PSS):NICU is a questionnaire assessing parents' feelings about their parenting role, exploring both positive aspects (e.g. emotional benefits, personal development) and negative aspects of parenthood (e.g. demands on resources, feelings of stress). Each item is graded on a Likert scale from 1-5, with responses coded as per published scoring instructions. Parental stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress.
Parent sense of competency (optional parent questionnaire) | Up to child's 2 years corrected age
  The Parent Sense of Competency Scale (PSOC) is a 17 item scale. Each item is rated on a 6 point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree". Several items on the PSOC are reverse coded as per poublished guidelines. A higher score indicates a higher parenting sense of competency. There are no average scores or 'cut-off's' for this tool.

CONTACTS AND LOCATIONS:
Overall Officials: Carmina Erdei, MD, Principal Investigator — Brigham and Women's Hospital and Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pineda R, Wallendorf M, Smith J. A pilot study demonstrating the impact of the supporting and enhancing NICU sensory experiences (SENSE) program on the mother and infant. Early Hum Dev. 2020 May;144:105000. doi: 10.1016/j.earlhumdev.2020.105000. Epub 2020 Mar 6. PMID 32151905
- [Background] Als H, Duffy FH, McAnulty GB, Rivkin MJ, Vajapeyam S, Mulkern RV, Warfield SK, Huppi PS, Butler SC, Conneman N, Fischer C, Eichenwald EC. Early experience alters brain function and structure. Pediatrics. 2004 Apr;113(4):846-57. doi: 10.1542/peds.113.4.846. PMID 15060237
- [Background] Pineda RG, Neil J, Dierker D, Smyser CD, Wallendorf M, Kidokoro H, Reynolds LC, Walker S, Rogers C, Mathur AM, Van Essen DC, Inder T. Alterations in brain structure and neurodevelopmental outcome in preterm infants hospitalized in different neonatal intensive care unit environments. J Pediatr. 2014 Jan;164(1):52-60.e2. doi: 10.1016/j.jpeds.2013.08.047. Epub 2013 Oct 17. PMID 24139564
- [Background] Pineda R, Raney M, Smith J. Supporting and enhancing NICU sensory experiences (SENSE): Defining developmentally-appropriate sensory exposures for high-risk infants. Early Hum Dev. 2019 Jun;133:29-35. doi: 10.1016/j.earlhumdev.2019.04.012. Epub 2019 May 1. PMID 31054467
- [Background] Thiim KR, Singh E, Mukundan S, Grant PE, Yang E, El-Dib M, Inder TE. Clinical experience with an in-NICU magnetic resonance imaging system. J Perinatol. 2022 Jul;42(7):873-879. doi: 10.1038/s41372-022-01387-5. Epub 2022 Apr 22. PMID 35459908
- [Background] Matthews LG, Walsh BH, Knutsen C, Neil JJ, Smyser CD, Rogers CE, Inder TE. Brain growth in the NICU: critical periods of tissue-specific expansion. Pediatr Res. 2018 May;83(5):976-981. doi: 10.1038/pr.2018.4. Epub 2018 Feb 7. PMID 29320484
- [Background] Dyet LE, Kennea N, Counsell SJ, Maalouf EF, Ajayi-Obe M, Duggan PJ, Harrison M, Allsop JM, Hajnal J, Herlihy AH, Edwards B, Laroche S, Cowan FM, Rutherford MA, Edwards AD. Natural history of brain lesions in extremely preterm infants studied with serial magnetic resonance imaging from birth and neurodevelopmental assessment. Pediatrics. 2006 Aug;118(2):536-48. doi: 10.1542/peds.2005-1866. PMID 16882805
- [Background] Kidokoro H, Anderson PJ, Doyle LW, Woodward LJ, Neil JJ, Inder TE. Brain injury and altered brain growth in preterm infants: predictors and prognosis. Pediatrics. 2014 Aug;134(2):e444-53. doi: 10.1542/peds.2013-2336. PMID 25070300